CLINICAL TRIAL: NCT03244501
Title: Modulation of Frontal Cortical Activity With Transcranial Static Magnetic Field Stimulation
Brief Title: Transcranial Static Magnetic Field Stimulation of Frontal Cortex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-1022
Record Dates: First submitted 2017-08-03; First posted 2017-08-09 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: tSMS; Transcranial Static Magnetic Field Stimulation; healthy control

STUDY DESIGN:
Intervention Model Description: All participants will receive three stimulations: left frontal, right frontal, and sham tSMS.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study, meaning that neither the participant nor the experimenter knows what kind of stimulation the participant is receiving. An unblinded monitor (separate from the staff that interacts with the participant) is responsible for providing the study coordinator with the active and sham magnet sequence. Each magnet has a number; the study coordinator is not aware which number corresponds to active or sham magnets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Left Frontal (Experimental): An active magnet (active tSMS) will be placed over the left frontal cortex, while a sham magnet (sham tSMS, a nonmagnetic metal cylinder made of brass) will be placed over the right frontal cortex.
  Interventions: Other: Active tSMS
- Right Frontal (Experimental): An active magnet (active tSMS) will be placed over the right frontal cortex, while a sham magnet (sham tSMS, a nonmagnetic metal cylinder made of brass) will be placed over the left frontal cortex.
  Interventions: Other: Active tSMS
- Sham Frontal (Sham Comparator): Sham magnets (sham tSMS, a nonmagnetic metal cylinder made of brass) will be placed over the left and right frontal cortex.
  Interventions: Other: Sham tSMS

INTERVENTIONS:
Other: Active tSMS — A cylindrical neodymium magnet is placed above the scalp.
  Arms: Left Frontal; Right Frontal
Other: Sham tSMS — A cylindrical piece of nonferrous metal (brass). This is not attracted to magnets, and is identical in weight and appearance to active magnets.
  Arms: Sham Frontal

SUMMARY:
The purpose of this study is to see if a new brain stimulation technique, static magnetic field stimulation (tSMS), which involves holding a static neodymium magnet over the scalp, can influence normal rhythms of brain activity.

DETAILED DESCRIPTION:
The investigator's primary objective is to determine the feasibility of modifying frontal brain activity using static magnetic fields. The investigator's will be examining the effects of static magnetic field of the spectral power of EEG data with healthy human participants.

This is a within-subjects design, where each participant will receive sham and active stimulation on the left and right frontal cortex. EEG data will be collected during each stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed, healthy, 18+ years old
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)
* Willing to comply with all study procedures and be available for the duration of the study - Speak and understand English

Exclusion Criteria:

* Medical history of Psychological/Emotional Disorders (depression, anxiety, bipolar, etc.)
* (For females) Pregnancy or breast feeding
* Diagnosis of eating disorder (current or within the past 6 months)
* Diagnosis of Obsessive-Compulsive Disorder (lifetime) Attention Deficit Hyperactivity Disorder (currently under treatment)
* Neurological disorders and conditions, including, but not limited to:
* History of epilepsy
* Seizures (except childhood febrile seizures and Electroconvulsive therapy-induced seizures)
* Dementia
* History of stroke
* Parkinson's disease
* Multiple sclerosis
* Cerebral aneurysm
* Brain tumors
* Medical or neurological illness or treatment for a medical disorder that could interfere with study participation (e.g., unstable cardiac disease, HIV/AIDS, malignancy, liver or renal impairment)
* Prior brain surgery Any brain devices/implants, including cochlear implants and aneurysm clips
* Any metal in/on the body, e.g., dental braces, glasses, piercings
* Traumatic brain injury
* Thick hair that would create distance between the magnet and the scalp
* Taking hormonal birth control or hormonal supplements (e.g., testosterone injections) - Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Electroencephalogram (EEG) Spectral Power | 4 minutes before stimulation, 10 minutes during stimulation, and 2 minutes after stimulation
  Changes in the spectral power of the EEG before (2 min eyes-closed, 2 min eyes-open), during (eyes-open), and after stimulation (eyes-open)

SECONDARY OUTCOMES:
Heart Rate Variability | 4 minutes before stimulation, 10 minutes during stimulation, and 2 minutes after stimulation
  Change in the ratio between the power in low frequency band and the power in high frequency band. As this outcome variable is a ratio between two items that are measured in microvolt^2, the ratio does not have a unit of measure.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States